CLINICAL TRIAL: NCT01055015
Title: A Randomized, Double-Blind, Study of the Analgesic Efficacy and Safety of Flexible Dose Q8003 Versus Low Dose Q8003 in Patients Who Have Undergone Primary Unilateral Total Knee Arthroplasty
Brief Title: Double Blind Efficacy and Safety Study of Flexible-Dose vs Low-Dose Q8003 After Undergoing Primary Unilateral Total Knee Arthroplasty
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: QRxPharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Q8003-009
Record Dates: First submitted 2010-01-22; First posted 2010-01-25 (Estimated); Last update posted 2012-05-17 (Estimated); Status verified 2012-05

CONDITIONS: Postoperative Pain
Keywords: total knee arthroplasty
MeSH Terms: conditions — Pain, Postoperative | interventions — Morphine; Oxycodone; MoxDuo

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Q8003, Flexible dose
  Interventions: Drug: Flexible dose Q8003 (morphine sulfate and oxycodone hydrochloride)
- 2 (Experimental): Q8003, Low dose
  Interventions: Drug: Low dose Q8003 (morphine sulfate and oxycodone hydrochloride)

INTERVENTIONS:
Drug: Flexible dose Q8003 (morphine sulfate and oxycodone hydrochloride) — IR Capsules, flexible dose, every 4 to 6 hours
  Arms: 1
Drug: Low dose Q8003 (morphine sulfate and oxycodone hydrochloride) — One 3 mg/2 mg IR Capsule every 4 to 6 hours following a 6 mg/4 mg loading dose.
  Arms: 2

SUMMARY:
This is a Phase 3, two-arm, double-blind study of efficacy and safety of Q8003 in patients who have undergone primary unilateral total knee arthroplasty

DETAILED DESCRIPTION:
This Phase 3 study is a two-arm, double-blind study to:

* compare the analgesic efficacy and safety of the flexible regimen of Q8003 (6 mg/4 mg up to 24 mg/16 mg) administered every 4-6 hours over a 48-hour Treatment Period versus low dose Q8003 (every 4-6 hours 3 mg/2 mg with a 6 mg/4 mg loading dose) to inpatients with moderate to severe postoperative pain who have undergone primary unilateral total knee arthroplasty.
* to evaluate the efficacy and safety of Q8003 when administered in the Voluntary Extension Period starting at 48 hours after the initial dosing and extending up to Day 12.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age at time of enrollment.
* If female, be at least one year post-menopausal, surgically sterile or practicing effective contraceptive, be non-lactating, and if of child-bearing potential, have a negative urine pregnancy test result.
* Have a body mass index (BMI) of 38 kg/m2 or less.
* Have undergone a primary unilateral total knee arthroplasty performed under under standardized general, spinal or epidural anesthesia.
* Have developed moderate to severe pain (a score of 2 or more on the 4 point Likert scale and at least 4 on the 11 point NPRS scale within 6 hours of discontinuing PCA on the morning after surgery).

Exclusion Criteria:

* In the opinion of the Investigator, has a history of pulmonary, cardiovascular (including uncontrolled hypertension), neurologic, endocrine, hepatic, gastrointestinal, or kidney disease or therapy that, in the opinion of the Investigator, would jeopardize the patient's well being by participation in this study or is mentally or emotionally unsuitable to participate, or unable/unwilling to comply with the study assessments.
* Used opiates continuously (including tramadol) for more than ten days in the past year.
* Hypersensitivity or poor tolerance to ibuprofen or short term opioids.
* Currently receiving any medications that are not at a stable dose (the same dose for > 2 months prior to date of surgery).
* Was dosed with another investigational drug within 30 days prior to the Screening Visit or has previously received treatment with Q8003.
* Current therapy with central nervous system depressant medications that might increase the risks of treatment with opioids (other than those used with surgical anesthesia).
* Current evidence of alcohol abuse (regularly drinks more than 4 units of alcohol per day; 1 unit = ½ pint of beer, 1 glass of wine, or 1 ounce of spirit).
* History of abusing licit or illicit drug substances within five (5) years of study entry.
* Has taken drugs known to interact with morphine or oxycodone metabolism, including, but not limited to, phenothiazines, monoamine oxidase inhibitors (MAOI), amphetamines, and muscle relaxants within the 4 weeks prior to the date of surgery.
* History of sleep apnea.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2010-02; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Difference in pain intensity scores from baseline | 48 hours

SECONDARY OUTCOMES:
Safety: adverse events, opioid-related signs and symptoms | Throughout the 48-hour period and during the voluntary safety extension period.

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Investigator Site, Birmingham, Alabama
  - Investigator Site, Sheffield, Alabama
  - Investigator Site, Phoenix, Arizona
  - Investigator Site, Laguna Hills, California
  - Investigator Site, Long Beach, California
  - Investigator Site, Pasadena, California
  - Investigator Site, Englewood, Colorado
  - Investigator Site, Edgewater, Florida
  - Investigator Site, Miami, Florida
  - Investigator Site, Sarasota, Florida
  - Investigator Site, Houston, Texas